CLINICAL TRIAL: NCT03647514
Title: A Prospective, Single-Arm Study to Evaluate the Efficacy and Safety of Abraxane Combined With Xeloda as Neo-Adjuvant Chemotherapy in Early Operable Breast Cancer
Brief Title: Abraxane Combined With Xeloda as Neo-Adjuvant Chemotherapy in Early Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: dingxwyh01
Record Dates: First submitted 2018-06-10; First posted 2018-08-27 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: neoadjuvant chemotherapy; Abraxane; Xeloda
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abraxane Combined With Xeloda (Experimental): Tailored neoadjuvant chemotherapy with 4 cycles of PX(weekly Abraxane 125mg/m2, Q3week Xeloda 1250mg/m2, 21day/cycle) is planned for early breast cancer patients(stage of T2-4N0-3M0) who are eligible for primary systemic therapy.
  Interventions: Drug: Abraxane; Drug: Xeloda

INTERVENTIONS:
Drug: Abraxane — Tailored neoadjuvant chemotherapy with 4 cycles of PX(weekly Abraxane 125mg/m2, Q3week Xeloda 1250mg/m2, 21day/cycle) is planned for early breast cancer patients(stage of T2-4N0-3M0) who are eligible for primary systemic therapy.
Drug: Xeloda — Tailored neoadjuvant chemotherapy with 4 cycles of PX(weekly Abraxane 125mg/m2, Q3week Xeloda 1250mg/m2, 21day/cycle) is planned for early breast cancer patients(stage of T2-4N0-3M0) who are eligible for primary systemic therapy.

SUMMARY:
Some studies have demonstrated the efficacy of Abraxane in treating breast cancer in both adjuvant and metastatic settings. Few data is available on Abraxane in neoadjuvant treatment for breast cancer.

The aim of this project is to evaluate tailored primary systemic therapy with weekly Abraxane (125mg/m2) Combined With Q3week Xeloda (1250mg/m2) in early operable (stage of T2-4N0-3M0) breast cancer. This study will be an open label non randomized, single arm, single center study.

DETAILED DESCRIPTION:
The hypothesis is that tailored neoadjuvant chemotherapy with 4 cycles of PX(weekly Abraxane 125mg/m2, Q3week Xeloda 1250mg/m2, 21day/cycle) is feasible and achieves high response rates.

It is proposed that 50 patients will be enrolled in this study. The target population is women with early breast cancer (stage of T2-4N0-3M0) who are eligible for primary systemic therapy.

The primary objective of the trial is to determine the overall response rate. Secondary endpoints will include response rates in axillary lymph nodes, safety and tolerability and the rate of breast conservation.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Women and men at least 18 years of age or older.
3. Pathological confirmation of breast cancer
4. Tumor stage(TNM):T2-4N0-3M0
5. No evidence of distant metastasis
6. Adequate bone marrow, hepatic, and renal function
7. Measurable disease as per RECIST criteria
8. Karnofsky≥70
9. Laboratory criteria:

PLT≥100*109/L WBC≥4000/mm3 HGB≥10g/dl ALT and AST<2*ULN

Exclusion Criteria:

1. Presence of metastatic disease.
2. Inflammatory breast cancer.
3. Bilateral breast cancer.
4. previous chemotherapy or hormonal therapy for current breast neoplasm.
5. other malignant tumors (concurrent or previous).
6. Pregnant woman.
7. Hypersensitive to any drug in Abraxane or Xeloda regimen or any ingredient of Abraxane or Xeloda.
8. Any severe systemic disease contraindicating chemotherapy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
ORR(CR+PR) | Following the completion of 12 weeks of neoadjuvant chemotherapy Treatment
  To evaluate the efficacy of concurrent Abraxane and Xeloda as neoadjuvant regimen in terms of: ORR(CR+PR), downstaging rates in tumor size and axillary lymph node.
  Pathological Complete Response(pCR) defined by: defined as ypT0, ypN0 (the absence of residual invasive and in situ cancer on evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy).

SECONDARY OUTCOMES:
Side Effects. | First Dose of Abraxane and Xeloda up to 24 months
  Determine side effects of these drugs like cardiotoxicity ,hematological toxicity，gastrointestinal symptoms and so on.
Event Free Survival(DFS) | Time of Surgery up to 5 years
  Time of surgery to first documentation of local or distant recurrence, or death or initiation of antineoplastic therapy before documentation of first relapse.
Overall Survival(OS) | First Dose of Abraxane and Xeloda up to 5 years
  Time from the first dose of Abraxane and Xeloda to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ding Xiaowen, Doc, Principal Investigator — Zhejiang Cancer Hospital

IPD SHARING:
Plan to Share IPD: No